CLINICAL TRIAL: NCT00830713
Title: Safety and Efficacy of Melanocyte-keratinocyte Transplantation in the Treatment of Vitiligo
Brief Title: Vitiligo Skin Transplantation
Acronym: MKTP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Iltefat Hamzavi, Dermatologist, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5385
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2010-05

CONDITIONS: Vitiligo
Keywords: vitiligo; skin transplantation; non-cultured; melanocyte; surgery
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MKTP treatment (Experimental): subject will undergo MKTP
  Interventions: Procedure: Melanocyte-keratinocyte transplantation procedure (MKTP)

INTERVENTIONS:
Procedure: Melanocyte-keratinocyte transplantation procedure (MKTP) — skin pigment cells are taken from areas of normal skin and placed on areas of that same person's body which have lost their color.

SUMMARY:
In vitiligo, the melanocytes are lost from the skin in certain areas. One treatment for vitiligo takes the melanocytes from areas of normal skin and places them on areas of that same person's body which have lost their color. This is called the melanocyte-keratinocyte transplantation procedure (MKTP). This procedure has been used successfully in over 3000 cases in India and Saudi Arabia. The purpose of this study is to see if it is effective when performed at the investigators' institution.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years old
2. Have a diagnosis of vitiligo with no news lesions or growth of old lesions in the past 6 months
3. Be able to understand the requirements of the study, the risks involved, and be able to sign the informed consent form
4. Agree to follow and undergo all study-related procedures

Exclusion Criteria:

1. Female patients who are breastfeeding, pregnant, or planning to become pregnant
2. Patients with a history of developing vitiligo or keloids at sites of trauma
3. Patients self-reported as having HIV or Hepatitis C
4. Patients self-reported as having uncontrolled Diabetes Mellitus
5. The investigator feels the patient should not participate in the study for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
effectiveness of MKTP in treating vitiligo | 6 months
  Assessed by percent repigmentation (excellent= 100%-95%, good= 94%-65%, fair= 64%-25%, poor= 24%-0%).

SECONDARY OUTCOMES:
safety of MKTP in treating vitiligo | 6 months
  Assessed by frequency of adverse events, including, scarring, infection, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Iltefat H Hamzavi, MD, Principal Investigator — Henry Ford Health Systems Dermatology Department
Locations (1):
- Henry Ford Medical Center, New Center One, Detroit, Michigan, United States

REFERENCES:
- [Background] Mulekar SV. Long-term follow-up study of segmental and focal vitiligo treated by autologous, noncultured melanocyte-keratinocyte cell transplantation. Arch Dermatol. 2004 Oct;140(10):1211-5. doi: 10.1001/archderm.140.10.1211. PMID 15492183
- [Background] Mulekar SV. Long-term follow-up study of 142 patients with vitiligo vulgaris treated by autologous, non-cultured melanocyte-keratinocyte cell transplantation. Int J Dermatol. 2005 Oct;44(10):841-5. doi: 10.1111/j.1365-4632.2005.02226.x. PMID 16207186